CLINICAL TRIAL: NCT06067321
Title: Comparison of Gastric Residual Volumes in Infants Fed at 4 and 6 Hours Prior to General Anaesthesia: A Randomised Controlled Trial
Brief Title: Gastric Residual Volumes in Infants Fed at 4 and 6 Hours Prior to General Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 334555
Record Dates: First submitted 2023-09-14; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Fasting; Anesthesia; Pediatric ALL
Keywords: gastric; volume
MeSH Terms: conditions — Fasting; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 hours formula feed (Active Comparator): Parents asked to offer formula feed 4 hours prior to anticipated procedure start
  Interventions: Other: abdominal ultrasound, insertion of naso-gastric tube
- 6 hour formula feed (Active Comparator): Parents asked to offer formula 6 hours prior to anticipated procedure start
  Interventions: Other: abdominal ultrasound, insertion of naso-gastric tube

INTERVENTIONS:
Other: abdominal ultrasound, insertion of naso-gastric tube — measurement antral cross sectional area, volume and pH of residual stomach contents

SUMMARY:
The safety implications of prolonged fasting in young children prior to general anaesthesia are well described. Current UK guidance recommends a fasting time of 6 hours for formula milk prior to general anaesthesia. European guidance published in 2022 recommended a reduced fast of 4 hours for infants taking formula milk, albeit with a downgraded level 2B of evidence given the paucity of high quality research in this area. Although pulmonary aspiration of gastric contents under anaesthesia in children is a rare event, animal studies suggest that aspiration of particulate matter at volumes greater than 0.8 ml/kg gastric volume are associated with demonstrable lung injury and mortality. Although rate of gastric emptying of formula preparations has been extensively studied in neonatal intensive care settings for preterm babies using ultrasound, few studies have measured gastric volume directly in healthy term infants undergoing anaesthesia.

DETAILED DESCRIPTION:
Traditional fasting guidelines of 6 hours for formula milk may be unnecessarily long. In practice, children also tend to be fasted for longer than the guidelines advise, as they may not always feed on cue, and delays in the hospital can occur on the day of surgery. Prolonged fasting in young children and infants is less well tolerated than in adults and can lead to hunger, dehydration and low blood sugar, as well as distress for the child and parents. We know from previous research in smaller babies that after a formula feed, the stomach empties by half in around 80 minutes, and empties completely by around 3 hours.

The investigators want to find out if young children and infants who are fed with formula milk 4 hours prior to an anaesthetic have similar levels of stomach contents at the time of their anaesthetic as those who are fed at 6 hours.

The investigators will carry out a clinical trial where children are randomised into 2 groups. Parents of children in Group 1 will be asked to offer a formula feed to their child 6 hours prior to the planned start time of their anaesthetic. Parents of children in Group 2 will be asked to offer a formula feed to their child 4 hours prior to the planned start time of their anaesthetic. Prior to having their anaesthetic a study team member will perform an abdominal ultrasound scan to check and record antral cross sectional area. Once asleep, gastric aspiration will be performed via naso-gastric tube. Volume, colour and pH of the fluid will be measure

The volume and acidity of any stomach contents will be compared between group 1 and group 2.

ELIGIBILITY:
Inclusion Criteria:

Term or term corrected (> 37 weeks) upto 12 months Formula fed ASA 1-3

Exclusion Criteria:

Significant reflux Co-administration of drugs known to impact gastric motility or PH of gastric contents Significant respiratory comorbidity including chronic lung disease on home oxygen Significant cardiac comorbidity

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
gastric residual volume | following induction, pre surgery
  aspiration of gastric contents via naso-gastric tube

SECONDARY OUTCOMES:
antral cross sectional area | pre induction
  ultrasound of abdomen

CONTACTS AND LOCATIONS:
Locations (1):
- Emily Saffer, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No